CLINICAL TRIAL: NCT07372391
Title: Effects of Janda's Approach Versus Instrument Assisted Soft Tissue Mobilization on Pain, Fatigue and Posture Among Individuals With Upper Cross Syndrome
Brief Title: Comparative Effects of Janda and IASTM on UCS
Acronym: IASTM UCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Dr. Khizra Hamid, Senior Lecturer, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPT/ERB/36; U1111-1334-3140 (Registry Identifier: WHO Universal Trial Number)
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Upper Cross Syndrome
Keywords: Janda's Approach; Instrument Assisted Soft Tissue Mobilization (IASTM); Upper Cross Syndrome (UCS); Pain; Fatigue; Posture
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus; Pain; Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Janda Group (Experimental): Participants in this arm received Janda's Approach that specifically targets functional muscular imbalance through stretching, strengthening and sensorimotor training.
  Interventions: Other: Janda's Approach
- IASTM Group (Active Comparator): Participants in this arm received Instrument Assisted Soft Tissue Mobilization through graston tool.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization (IASTM)

INTERVENTIONS:
Other: Janda's Approach — All programs will be performed 3 times per week for 4 weeks. Each session will be of 45 minutes. 15 minutes warm up, 10 minutes cool down with 20 minutes stretching and isometrics along with sensorimotor training. Static stretching will be performed holding the stretch for at least 15 sec. and isometric exercise will be conducted three times in a maximum contraction mode for 3 sec under the supervision of a certified expert. Sensorimotor training includes following tasks chin tuck ins, scapular setting, wall alignment drills, diagonal arm patterns.
  Arms: Janda Group
Other: Instrument Assisted Soft Tissue Mobilization (IASTM) — It will be performed 3 times per week for 4 weeks. Each treatment session will be of 45 minutes. 15 minutes Warm up and 10 minutes cool down period and 20 mins application of IASTM assisted by gel or oil to make it friction free. Icing will be applied at end of each session to reduce post treatment inflammation.
  Arms: IASTM Group

SUMMARY:
Upper Crossed Syndrome (UCS) is a widespread muscle imbalance defined by tightness in the upper trapezius, pectoralis major and minor, and sternocleidomastoid, coupled with weakness in deep neck flexors, lower trapezius, and serratus anterior. It is usually triggered by sustained faulty posture, predominantly in computer users, drivers, or other prolonged forward head and trunk flexion positions, resulting in pain, fatigue, limited ROM and functional limitations.

On a global scale, estimates suggest that UCS affects between 11% and 60% of individuals, spanning various age groups and cultural backgrounds. Individuals who engage in prolonged slouching, such as desk workers, teachers, drivers, IT professionals, students, and laundry workers, demonstrate prevalence rates of approximately 32.4%, 16.2%, 26.4%, 67%, 37.1%, and 28% respectively.

Janda's approach, aims to restore or normalize muscle balance and refine posture by combining stretching of tight and overactive muscles with strengthening of weak and inhibited muscles, in sequence. Instrument-Assisted Soft Tissue Mobilization (IASTM) enhances ROM and alleviates pain by directing myofascial restrictions. As adjuncts, hot packs and transcutaneous electrical nerve stimulation (TENS) are frequently used to reduce discomfort and prepare tissues for further therapeutic interventions.

Although numerous intervention techniques are offered for UCS but limited research has compared Janda's approach and IASTM, especially with respect to their impact on fatigue. Therefore, this study aims to evaluate and compare the effects of these interventions on pain, fatigue, and posture in adults with UCS.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 19-44 years (Adults), both genders
* Pectoralis major and Upper trapezius tightness, Serratus anterior and Lower trapezius weakness
* Forward Head Posture (developed within 6 weeks or more than 3 months)
* Reported neck, upper back, or shoulder pain or discomfort
* Pain 5 or above on NPRS for at least 3 months
* Fatigue score of 4 or above on Fatigue Severity Scale

Exclusion Criteria:

* Congenital anomalies
* Thoracic Outlet Syndrome
* Inflammatory disorders
* Headache due to any cause (migraine, disc bulge)
* Postural defects (Torticollis, Scoliosis)
* Malignancy
* Fracture of cervical spine and clavicle

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Baseline, Post-intervention 2 weeks, Post-intervention 4 weeks
  Pain intensity measured using the Numeric Pain Rating Scale (NPRS), an 11-point scale rating from 0 (no pain) to 10 (worst pain).
Fatigue | Baseline, Post-intervention 2 weeks, Post-intervention 4 weeks
  Fatigue assessed using the Fatigue Severity Scale (FSS), a 9-item self-report questionnaire in which each item is scored on a 7-point Likert scale, with higher scores indicating greater fatigue severity.
Posture | Baseline, Post-intervention 2 weeks, Post-intervention 4 weeks
  REEDCO Posture Assessment Scale was employed to evaluate postural alignment in individuals with Upper Crossed Syndrome, focusing specifically on the head, shoulder, and upper back regions. These items were selected as they directly correspond to the primary postural deviations associated with the syndrome, namely forward head posture, rounded shoulders, and increased thoracic kyphosis. Scoring was based on established REEDCO criteria, a score of 10 (normal alignment or good posture), a score of 5 (minimal to moderate deviation or fair posture), and a score of 0 (marked or severe deviation or poor posture)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Biological and Applied Sciences, Lahore, Lahore, Punjab Province, Pakistan